CLINICAL TRIAL: NCT05545683
Title: Open-Label Phase 3 Clinical Study to Investigate Safety and Immunogenicity of a Single VLA2001 Booster Vaccination in Volunteers Aged ≥18 Years, After Priming With Another Inactivated COVID-19 Vaccine
Brief Title: Safety and Immunogenicity of Inactivated Heterologous Booster Vaccination
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: funding was suspended
Sponsor: Centro de Estudios en Infectogía Pediatrica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT-VAL-LOP-COV-001
Record Dates: First submitted 2022-09-06; First posted 2022-09-19 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VLA 2001 (Experimental): One dose (0.5 mL) contains no less than 25 Antigen Units (AU) of inactivated SARS-CoV-2.
  Highly purified whole virus SARS-CoV-2 antigen, inactivated and adjuvanted with CpG 1018 in combination with aluminum hydroxide.
  Interventions: Biological: VLA 2001

INTERVENTIONS:
Biological: VLA 2001 — VLA2001 is a highly purified whole virus, inactivated, adjuvanted vaccine, using the manufacturing platform of Valneva's encephalitis (JE) vaccine

SUMMARY:
Data from some studies indicate the decline in the effectiveness of the authorized COVID-19 vaccines due to antibody waning following vaccination and the emergence of different variants. These findings support the need to increase vaccination and booster campaigns to protect the adult population against infection. Valneva developed the VLA2001 vaccine, a highly purified, whole virus SARS-CoV-2 vaccine produced on Vero cells and inactivated with β-propiolactone. VLA2001 will be adjuvanted with the licensed adjuvant cytosine phospho-guanine (CpG) 1018 (produced by Dynavax, contained in HEPLISAV-B®) in combination with aluminum hydroxide. On April 14, 2022, VLA2001 was granted Conditional Marketing Authorization (CMA) by the Medicines and Healthcare products Regulatory Agency (MHRA) of the United Kingdom for primary immunization in adults 18 to 50 years of age. This follows the emergency use authorization granted by the Bahraini NHRA in March 2022. As a substantial population has received a primary vaccination series with authorized vaccines, a booster dose to extend the duration and protection may be required.This study aims to investigate the safety, tolerability, and immunogenicity of the VLA2001 vaccine as a booster dose to adults 18 years and older who were primed with another licensed inactivated COVID-19 vaccine at least 6 months prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of either gender aged 18 years and older at screening
2. Participants who have received two doses of an inactivated Covid vaccine and no booster. Primary series with an inactivated vaccine had to be completed at least 6 months prior to enrollment.
3. Participants must have read, understood, and signed the informed consent form (ICF)
4. Medically stable such that, according to the judgment of the investigator, hospitalization within the study period is not anticipated and the participant appears likely to be able to remain on study through the end of protocol-specified follow-up.

   a. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to the expected day of booster vaccination.
5. Participant has a Body Mass Index (BMI) of 18.0-30.0 kg/m2, inclusive, at screening (Visit 0).
6. Must be able to attend all visits of the study and comply with all study procedures, including daily completion of the e-diary for 7 days following each vaccination.
7. Women of childbearing potential (WOCBP), who are sexually active with a man, must be able and willing to use at least 1 highly effective method of contraception (i.e. implant contraceptive, intra-uterine device (IUD) containing either copper or levonorgestrel, male sterilization [vasectomy], female sterilization, injectable contraceptive, oral contraceptive pill, vaginal contraceptive ring, barrier type of birth control measure) from study start until a minimum of 3 months after receiving the booster vaccine.

   1. A female participant is considered to be a WOCBP after menarche and until she is in a postmenopausal state for 12 consecutive months (without an alternative medical cause) or otherwise permanently sterile.
   2. Note: Participants not of childbearing potential are not required to use any other forms of contraception during the study. Non-childbearing potential is defined as participant confirmed:
   3. Surgical sterilization for ≥3 months prior to Visit 1 (e.g., bilateral oophorectomy, bilateral salpingectomy, bilateral occlusion by cautery, hysterectomy, or tubal ligation).
   4. Postmenopausal (defined as permanent cessation of menstruation for at least 12 consecutive months prior to screening).
8. WOCBPs must have a negative pregnancy test prior to the booster vaccination.
9. Has received a second dose of licensed inactivated COVID-19 vaccine 6 to 15 months before study vaccination.

Exclusion Criteria:

1. Known history of natural SARS-CoV-2 infection (based on medical history and/or confirmed either by PCR or rapid antigen test) less than four months prior to the planned booster vaccination..
2. Participant is pregnant or planning to become pregnant within 3 months after booster administration.
3. History of allergy to any component of the vaccine.
4. Participant had close contact to persons with confirmed SARS-CoV-2 infection within 30 days prior to screening (Visit 0).
5. Participant has participated in a clinical study involving an investigational SARS-CoV-2 vaccine or has received or plans to receive a licensed SARS-CoV-2 vaccine during the duration of the study.
6. Significant infection or other acute illness, including fever > 100 °F (> 37.8 °C) within 48 hours before vaccination.
7. Positive SARS-CoV-2 rapid Antigen test result during screening (Visit 0) or Visit 1.
8. Participant has a known or suspected defect of the immune system, such as participants with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to the expected day of vaccination (Visit 1).

   * Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent ≥ 0.05 mg/kg/day within 4 weeks prior to the expected day of first vaccination (visit 1), radiation therapy or immunosuppressive cytotoxic drugs/ monoclonal antibodies in the previous 3 years; topical and inhaled steroids are allowed.
   * Participants with chronic HIV unless: HIV disease with documented viral load <50 copies/ml and CD4 count >200 cells/mm3 for at least 6 months before first vaccination, and stable antiretroviral therapy for the last 6 months.
9. Participant has a history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than 5 years ago that is considered to have achieved a cure, the participant may be enrolled. A history of hematologic malignancy is a permanent exclusion. Participants with a history of skin cancer must not be vaccinated at the previous tumor site.
10. History of drug dependency or current use of drug of abuse or alcohol abuse at screening.
11. Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to the expected day of first vaccination (Visit 1).
12. History of clinically significant bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
13. Severe and uncontrolled ongoing autoimmune or inflammatory disease, History of Guillain-Barre syndrome or any other demyelinating condition.
14. Any other significant disease, disorder or finding which in the opinion of the investigator may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
GMT fold-rise for neutralizing antibodies D1 and D16 | Day of vaccination (D1) and 15 days after vaccination (D16)
  GMT fold-rise for neutralizing antibodies against SARS-CoV-2 15 days after a single booster dose with VLA2001
Adverse events | From the day of vaccination (D1) until 7 days after vaccination (D8)
  Frequency and severity of solicited AEs (local and systemic reactions) after the VLA2001 booster vaccination

SECONDARY OUTCOMES:
Individual neutralizing antibody titers D1, D16, D181, M9, M12 | Day of vaccination (D1), 15 days after vaccination (D16), 180 after vaccination (D181), 9 months after vaccination (M9) and 12 months after vaccination (M12)
  Immune response as determined by the GMT of SARS-CoV-2-specific neutralizing antibodies
GMT fold-rise for neutralizing antibodies D1, D181, M9, M12 | 180 after vaccination (D181), 9 months after vaccination (M9) and 12 months after vaccination (M12)
  GMT fold-rise for neutralizing antibodies against SARS-CoV-2 following a single booster dose with VLA2001.
Proportion of participants achieving fold rise in neutralizing antibodies D16, D181, M9, M12 | 15 days after vaccination (D16), 180 after vaccination (D181), 9 months after vaccination (M9) and 12 months after vaccination (M12)
  Proportion of participants achieving an at least 2-, 4-, 10- or 20-fold rise over baseline (pre-booster) in terms of neutralizing antibodies to SARS-CoV-2 S-protein
GMT fold-rise of IgG antibodies D1, D16, D181, M9, M12 | Day of vaccination (D1), 15 days after vaccination (D16), 180 after vaccination (D181), 9 months after vaccination (M9) and 12 months after vaccination (M12)
  GMT fold-rise of IgG antibodies to the SARS-CoV-2 S-protein following a single booster dose with VLA2001.
GMT of IgG antibodies to the SARS-CoV-2 S-protein D1, D16, D181, M9, M12 | Day of vaccination (D1), 15 days after vaccination (D16), 180 after vaccination (D181), 9 months after vaccination (M9) and 12 months after vaccination (M12)
  Immune response as determined by the GMT of IgG antibodies to the SARS-CoV-2 S-protein
Fold-rise IgG antibodies to SARS-CoV-2 S-protein D16, D181, M9, M12 | 15 months after vaccination (D16), 180 after vaccination (D181), 9 months after vaccination (M9) and 12 months after vaccination (M12)
  Proportion of participants achieving an at least 2-, 4-, 10- or 20-fold rise over baseline (pre-booster) in terms of IgG antibodies to SARS-CoV-2 S-protein
T-cell response | From the day of vaccination (D1) until month 12 after vaccination day
  Assessment of T-cell responses from PBMCs in a subset of participants after in vitro stimulation with SARS-CoV-2 antigens using e.g. ELISpot (IFN γ) or intracellular cytokine staining (IL-2, IL-4, IL-5, IL-13, TNFα, IFN γ)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Lopez-Medina, MD, Principal Investigator — Scientific Director
Locations (1):
- Centro de Estudios en Infectología Pediátrica, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No